CLINICAL TRIAL: NCT01443234
Title: OxIGen: Oxford Imagery Generation: Investigating the Effects of an Internet Based Computer Program in Depression
Acronym: OxIGen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Lupina Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11/SC/0278
Record Dates: First submitted 2011-09-27; First posted 2011-09-29 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2013-06

CONDITIONS: Depression
Keywords: Depression; Cognitive Bias; Internet
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- OxIGen program (Experimental): Internet based intervention taking place over 4 weeks
  Interventions: Other: OxIGen
- OxIGen: control version (Placebo Comparator): A control version of the internet-based OxIGen intervention
  Interventions: Other: OxIGen: control version

INTERVENTIONS:
Other: OxIGen — Internet-based intervention with 12 sessions over 4 weeks
  Arms: OxIGen program
Other: OxIGen: control version — A control version of the OxIGen internet-based intervention (i.e. identical but with putative active components removed)
  Arms: OxIGen: control version

SUMMARY:
This research study is designed to investigate the effects of an online computer program, called OxIGen (Oxford Imagery Generation), on thinking style and mood in depression. The OxIGen program will be delivered online over four weeks and with follow-up at one, three and six months. This will inform potential future development of this computerized task into an online intervention to modify negative thinking styles in depression.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give consent to the study
* Male or Female, aged between 18 and 65 years
* Current Major Depressive Episode (assessed by semi-structured clinical interview)
* Access to internet in order to complete the online program
* Able to travel to research centre for assessment appointments
* Fluent in written and spoken English

Exclusion Criteria:

* Meets criteria for current psychotic disorder
* History of mania or hypomania as assessed by semi-structured clinical interview, or has elsewhere received a diagnosis of Bipolar disorder
* Antidepressant medication begun or changed in dosage during last month
* Meets criteria for current substance abuse disorder
* Involved in other current treatment trials
* Currently receiving psychological therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-02; Primary Completion 2013-04 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in score on Beck Depression Inventory - II | Baseline and post-intervention (4 weeks)

SECONDARY OUTCOMES:
Change in score on Quick Inventory of Depressive Symptoms - Self Report | Baseline and post-intervention (4 weeks)
Change in State-Trait Anxiety Inventory (Trait scale) | Baseline and Post-Intervention (4 weeks)
Change on Beck Anxiety Inventory | Baseline and Post-Intervention (4 weeks)
Change on Scrambled Sentences Task | Baseline and Post-Intervention (4 weeks)
Change on Life Orientation Test - Revised | Baseline and Post-Intervention (4 weeks)
Change on Prospective Imagery Test | Baseline and Post-Intervention (4 weeks)
Change on Behavioural Activation in Depression Scale | Baseline and Post-Intervention (4 weeks)
Change in IAPT Toolkit | Baseline and Post-Intervention (4 weeks)
  Includes the GAD-7, PHQ-9 and Work and Social Adjustment Scale
Change on EuroQol-5D | Baseline and Post-Intervention (4 weeks)
Change in Neuroticism | Baseline and Post-Intervention (4 weeks)
Change on Beck Depression Inventory - II | Baseline and Follow-Up (one month, three months, six months)
Change on Quick Inventory of Depressive Symptoms - Self Report | Baseline and Follow-Up (one month, three months, six months)
Change on State-Trait Anxiety Inventory (Trait scale) | Baseline and Follow-Up (one month, three months, six months)
Change on Beck Anxiety Inventory | Baseline and Follow-Up (one month, three months, six months)
Change on Life Orientation Test - Revised | Baseline and Follow-Up (one month, three months, six months)
Change on Prospective Imagery Test | Baseline and Follow-Up (one month, three months, six months)
Change on Behavioural Activation in Depression Scale | Baseline and Follow-Up (one month, three months, six months)
Change on IAPT Toolkit | Baseline and Follow-Up (one month, three months, six months)
  Includes GAD-7, PHQ-9, Work and Social Adjustment Scale
Change on Euroqol-5D | Baseline and Follow-Up (one month, three months, six months)
Change on Neuroticism | Baseline and Follow-Up (one month, three months, six months)
Image Generation Task | Post-Intervention (4 weeks)
  Task adapted from Sharot et al. (2007, Nature)

CONTACTS AND LOCATIONS:
Overall Officials: Emily A Holmes, D.Clin.Psy, PhD, Principal Investigator — University of Oxford
Locations (2):
- United Kingdom (2):
  - MRC Cognition and Brain Sciences Unit, Cambridge, Cambridgeshire
  - Department of Psychiatry, University of Oxford, Oxford, Oxfordshire